CLINICAL TRIAL: NCT01776437
Title: A Phase 1 Food Effect Study of BMN 673 Administered to Healthy Adult Male Volunteers
Brief Title: Study of BMN 673, a PARP Inhibitor, in Healthy Adult Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 673-103
Record Dates: First submitted 2013-01-24; First posted 2013-01-28 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Human Volunteers
MeSH Terms: interventions — talazoparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A (Experimental): Period 1: fasted control → Period 2: fed control
  Interventions: Drug: BMN 673
- Treatment B (Experimental): Period 1: fed control → Period 2: fasted control
  Interventions: Drug: BMN 673

INTERVENTIONS:
Drug: BMN 673 — 500mcg dose of BMN 673, 2 discrete single doses separated by 21 days

SUMMARY:
This is a randomized, 2-period, 2-sequence crossover study to evaluate the effect of food on the relative bioavailability of BMN 673 during fasting and fed conditions in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male, between the ages of 18 and 55.
* Non-smoking for at least 1 year before Screening.
* Willing and able to provide informed consent.
* Have a BMI between 18 to 30kg/m2.
* Willing and able to comply all study procedures.
* Have adequate organ function
* Sexually active patients must be willing to use an acceptable method of contraception.

Exclusion Criteria:

* History of any illness that might confound the results of the study or pose an additional risk in administering study medication to the subject.
* Current use of prescription medication or regular treatment with over-the-counter medications.
* Consumption of herbal medications or dietary supplements.
* Consumption of more that than 3 units of alcoholic beverages per day.
* Consumption of more than five 240-mL servings of coffee or other caffeinated beverage.
* History of alcohol or drug abuse or addiction within 6 months of study entry.
* Participation in a clinical Study involving administration of an investigational drug within 1 month or 5 half lives (whichever is longer).
* Donation of any blood or having had a significant loss of blood with 56 days.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2013-02; Primary Completion 2013-05 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
The primary outcome of this study is to evaluate the effect of food on the relative bioavailability of BMN 673. The Pharmacokinetic analyses of plasma BMN 673 concentration-time will be measured using non-compartmental methods. | 4 months

SECONDARY OUTCOMES:
Assess the safety and tolerability of BMN 673 during fasting and fed conditions with the following safety assessments: adverse events, physical examination, vital signs, concomitant medications, clinical laboratory tests and ECG. | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Covance Clinical Research Unit Inc., Evansville, Indiana, United States